CLINICAL TRIAL: NCT03066973
Title: THE EFFECTIVENESS OF BREATHING EXERCISES TO LABOR PAIN and DURATION: A RANDOMIZED CONTROLLED TRIAL
Brief Title: BREATHING EXERCISES FOR LABOR PAIN AND DURATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Yasemin Cayir, Assoc. Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/69
Record Dates: First submitted 2017-02-21; First posted 2017-03-01 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Labor Pain; Breathing Exercise
Keywords: breath exercises; labor pain; labor duration; VAS
MeSH Terms: conditions — Labor Pain | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The trial compares nulliparous pregnant in the second stage of labor instructed regarding breathing exercise with a control group that received standard care service.
  Interventions: Behavioral: BREATHING EXERCISE
- Control group (No Intervention): control group that received standard care service.

INTERVENTIONS:
Behavioral: BREATHING EXERCISE — The intervention group was instructed on breathing exercise according to the established trial protocol.
  Arms: Intervention group

SUMMARY:
This study aimed to assess the efficacy of breathing exercises (BE) during the second stage of labor for maternal pain, duration of labor and first-minute APGAR score. This is a randomized controlled trial that compares nulliparous pregnant in the second stage of labor instructed regarding BE with a control group (CG) that received standard care service. It was conducted at Nenehatun Obstetric and Gynecology Hospital between May-June 2016, in Erzurum. One session of BE training were given to pregnant in intervention group (IG). Visual Analog Scale (VAS) was performed to identify perception of pain to all pregnant during the second stage of birth. Time of the second stage was recorded as second (sec), and first minute APGAR scores were recorded. Significance was set at p<0.05.

DETAILED DESCRIPTION:
In this trial, it is aimed to assess the effectiveness of breathing exercises (BE) for management of labor pain during the second stage of labor. Nulliparous pregnant were randomized two arms. Intervention group received breathing exercise at the first stage of labor. Control group received routine care services. It was conducted at Nenehatun Obstetric and Gynecology Hospital between May-June 2016, in Erzurum, Turkey. Visual Analog Scale (VAS) was performed to identify perception of pain to all pregnant during the second stage of labor. Time of the second stage was recorded as second (sec), and first minute APGAR scores of newborn were recorded. All analysis was carried out using SPSS 20. Significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Nullipar females
* Gestational age 37-42 week

Exclusion Criteria:

* Analgesic and anestezice use
* Clinical instability
* Psychiatric disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — nullipar females
Enrollment: 250 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Labor pain | 1 MONTH
  It will be measured by Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Duration of labor | 1 MONTH
  It will be measured at the second stage of labor as second.
APGAR score | 1 MONTH
  It will be measured by APGAR score by on-duty pediatrician during assesment at the birth room.

IPD SHARING:
Plan to Share IPD: Yes
it will be submitted as an article

REFERENCES:
- [Derived] Yuksel H, Cayir Y, Kosan Z, Tastan K. Effectiveness of breathing exercises during the second stage of labor on labor pain and duration: a randomized controlled trial. J Integr Med. 2017 Nov;15(6):456-461. doi: 10.1016/S2095-4964(17)60368-6. PMID 29103415